CLINICAL TRIAL: NCT06325644
Title: Feasibility and Efficacy of a Well-Formulated Ketogenic Diet in Delaying Progression of Polycystic Kidney Disease in Patients at Risk for Rapid Progression
Brief Title: Well-Formulated Ketogenic Diet Polycystic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023H0258; CDMRP-PR212399-G (Other Grant/Funding Number: Departent of Defense)
Record Dates: First submitted 2024-02-26; First posted 2024-03-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Diet, Ketogenic; Ketones; Blood Specimen Collection; Body Composition; Glomerular Filtration Rate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): The KD will follow general principles the investigators have described with the aim to achieve blood ketones >0.5 mM, which will require most participants to consume <50 g/day carbohydrate and ~1.5 g/kg reference weight protein. Fat will comprise the remaining calories with an emphasis on monounsaturated and saturated sources from whole foods.
  Interventions: Other: Ketogenic Diet; Biological: Ketone/Glucose Monitoring; Biological: CGM/CKM; Biological: Blood Draw; Other: Body Composition; Other: Change in glomerular filtration rate (mg/mmol) via magnetic resonance imaging (MRI) .

INTERVENTIONS:
Other: Ketogenic Diet — The diet intervention will start after all baseline testing is complete
Biological: Ketone/Glucose Monitoring — KetoMojo hand-held glucometer will be used daily to monitor dietary intervention adherence.
Biological: CGM/CKM — Continuous Ketone/Glucose Monitor will be applied at the start of Test Day 1. The sensor will be checked by the study team at each test day and will be removed and replaced by a fresh sensor at ~2- week intervals during the study. The sensor will be removed at the end of the final test day.
Biological: Blood Draw — Blood samples will be collected according to the schedule in Figure 1
Other: Body Composition — DEXA Scanning will be done pre-, mid-, and post- intervention.
Other: Change in glomerular filtration rate (mg/mmol) via magnetic resonance imaging (MRI) . — Changes in glomerular filtration rate will be assessed via magnetic resonance imagining conducted by trained professionals. MRI imaging analyses will determine cardiac function. Trained imaging professionals will analyze the images to determine overall change (mg/mmol).

SUMMARY:
This is a prospective study to determine ketogenic diet effect on htTKV, GFR, microalbuminuria. This is a single-center study of 20 patients with ADPKD and deemed high risk for progression to ESRD. This determined by combination of features of ADPKD and htTKV as assessed by prior computed tomography (CT) or MRI. Patients will be recruited from the Polycystic Kidney Disease (PKD) Clinic at Ohio State University Wexner Medical Center. Enrolled patients will have MRI for htTKV, urinary studies, blood tests at baseline, 6 months, and 52 weeks. Blood for GFR will be assessed three times over the course of the study including baseline, 6 months, and 1 year. Participants will follow ketogenic diet for 52 weeks. Investigatory diet team will manage the ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Diagnosis of ADPKD by imaging and/or genetic testing
* GFR ≥ 25 mg/dl
* Patients at risk for rapid progression of ADPKD: Mayo Class 1C-1E along with any other high risk features including early decline in GFR, hypertension onset ≤ 35 years of age, urologic events ≤ 35 years of age, PKD 1 truncating mutation and PROPKD score of 4 or higher as determined by the treating physician
* No changes of medications within the last three months.
* Able to comply with dietary intervention
* Ability to sign informed consent

Exclusion Criteria:

* Patients currently being treated with Tolvaptan
* Diagnosed with diabetes.
* Pregnancy
* Contraindications to MRI
* Ketogenic diet within the last three months
* Severe kidney disease with GFR < 25 mg/dl
* Unable to purchase food for the diet intervention
* Gastrointestinal disorders that will interfere with diet intervention
* Chronic alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Finger Stick Beta-Hydroxybutyrate | Up to ~ 52 Weeks
  changes in fasting ketone levels.
Finger Stick Glucose | Up to ~ 52 Weeks
  changes in fasting glucose levels.

SECONDARY OUTCOMES:
Blood Pressure | Time Frame: Up to ~ 12 Weeks
  Changes in both Systolic and Diastolic blood pressure will be measured at each lab visit (eg. Baseline, Week 6, and Week 12).
  Recording: The systolic and diastolic pressures are recorded in millimeters of mercury (mmHg). For example, a reading of "120/80 mmHg" indicates a systolic pressure of 120 mmHg and a diastolic pressure of 80 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-01-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT06325644/Prot_000.pdf
  • Informed Consent Form (2024-01-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT06325644/ICF_001.pdf